CLINICAL TRIAL: NCT00740142
Title: Efficacy of Combined Oral L-ornithine-L-aspartate and Oral Lactulose in Patients With Hepatic Encephalopathy
Brief Title: Efficacy of Combined Oral L-ornithine-L-aspartate and Lactulose in Patients With Hepatic Encephalopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si 341/2008
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Hepatic Encephalopathy
Keywords: L ornithine L aspartate; Lactulose; Hepatic encephalopathy; LOLA
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — ornithylaspartate; Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Interventional arm: oral L-ornithine-L-aspartate and oral lactulose
  Interventions: Drug: L-ornithine-L-aspartate and lactulose
- 2 (Placebo Comparator): Oral lactulose
  Interventions: Drug: placebo and lactulose

INTERVENTIONS:
Drug: L-ornithine-L-aspartate and lactulose — L-ornithine-L-aspartate 1 sachet(3 grams)3 times a day for 7 days
  Arms: 1
Drug: placebo and lactulose — placebo 3 times a day for 7 days
  Arms: 2

SUMMARY:
Hypothesis: Is the combination of oral L-ornithine-L-aspartate and lactulose more efficacious than oral lactulose alone in treatment of hepatic encephalopathy? Study design; Randomized, double-blinded, placebo controlled trial

DETAILED DESCRIPTION:
Data collection

1. Baseline characteristics

   * demographic data; age, gender, BW, height
   * cirrhosis; cause, duration, Child-Pugh score,complications of cirrhosis such as EV, ascites, hepatic encephalopathy, SBP etc.
   * comorbidity such as DM, CVA
2. After randomization

   * assessment of mental status (West-Haven criteria), Portal-systemic encephalopathy index (PSEI), number connection test, serum ammonia, asterixis at Day 1,3,7 and EEG at day 1,7
   * blood chemistry such as CBC, BUN, Creatinine, electrolyte, LFT, coagulogram, BS at Day 1,3,7
   * record adverse effect of drug such as nausea, vomiting, bloating.
   * record diet, frequency of bowel movement and stool pH
   * compliance

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Age 18-80
* Hepatic encephalopathy grade II-III
* Serum ammonia > 60 mcg/mL
* Informed consent

Exclusion Criteria:

* Recent GI hemorrhage
* Severe sepsis
* Degenerative CNS disease or major psychiatric illness
* Serum creatinine > 1.5 mg/dl
* Pregnancy or lactation
* Poorly controlled DM
* Insertion of TIPS
* Received CNS depressants or hypnotics
* Treatment with metronidazole, kanamycin or branched-chain amino acid
* Hypersensitivity to L-ornithine-L-aspartate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2010-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To assess improvement of mental status of the patients | 7 days

SECONDARY OUTCOMES:
To assess improvement of number connection test, serum ammonia, EEG, asterixis and PSE index of the patients | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Siwaporn Chainuvati, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok, Thailand